CLINICAL TRIAL: NCT00847470
Title: Reasons for Placing the First Restoration on Permanent Tooth Surfaces
Brief Title: DPBRN Reasons for Placing the First Restoration on Permanent Tooth Surfaces
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); University of Copenhagen (Other); University of Florida (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Gregg H. Gilbert, DDS, MBA, FAAHD, Gregg H. GIlbert, DDS, MBA, Study Chair, University of Alabama at Birmingham, Dental Practice-Based Research Network
Other Study IDs: 101883
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Dental Caries
Keywords: Dental caries; Assessments; dental materials
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to document the reasons for placing the first restoration ("filling") on a previously un-restored surface in a permanent ("adult") tooth.

DETAILED DESCRIPTION:
The aims of this study were to (1) quantify DPBRN practitioner-investigators pre-operative and post-operative assessments of the depth of the caries lesion being treated; (2) quantify the prevalence of dental material types used to restore the first restoration in a permanent tooth surface; and (3) test the hypothesis that DPBRN practitioner investigators in the "Assessment of caries diagnosis and caries treatment" study who stated that they wait until the caries lesions reach dentin before they place the first restoration are in fact more likely in this study to do restoration in teeth that have caries reaching into dentin.

The aims were met by enrolling 230 DPBRN practitioner-investigators in the "Reasons for placing the first restoration on permanent tooth surfaces" study, each of whom recorded information about approximately 50 consecutive restorations that they placed on unrestored surfaces. This study about restorative treatment received by patients provided the opportunity to record the variations in the treatment provided, and also provided a basis for subsequent future studies to investigate how defects on fillings develop over time. These results will also be related to the findings from "Assessment of caries diagnosis and caries treatment" study where practitioners outlined how they detected dental decay, the stage at which the decay was treated by placing fillings, and how they rely on preventive measures to stop the decay process without placing fillings.

ELIGIBILITY:
Inclusion Criteria:

* participants directly involved in this study were patients who sought dental treatment in the practitioner-investigators' practices
* any tooth surface that was previously unrestored was eligible for this study, provided that it was on a permanent ("adult") tooth. This means that permanent first molars were eligible, which typically erupt at about age 6 years. This means that persons age 6 and older were enrolled in the study and there was no upper age limit.

Exclusion Criteria:

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Practitioner investigators must have been enrolled in the DPBRN, completed the "Assessment of caries diagnosis & caries treatment" study; and do at least some restorative dentistry in their practices. The human subjects directly involved in this study were patients who had sought treatment in the DPBRN practitioners' practices.
Sampling Method: Probability Sample
Enrollment: 5810 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H. Gilbert, DDS, MBA, Study Chair — Dental Practice-Based Research Network; Valeria V. Gordan, DDS, MS, MSCI, Principal Investigator — Dental Practice-Based Research Network
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- [Derived] Litaker MS, Gordan VV, Rindal DB, Fellows JL, Gilbert GH; National Dental PBRN Collaborative Group. Cluster Effects in a National Dental PBRN restorative study. J Dent Res. 2013 Sep;92(9):782-7. doi: 10.1177/0022034513497752. Epub 2013 Jul 15. PMID 23857643
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org
- See also: Dental Practice-Based Research Network — http://DPBRN.org